CLINICAL TRIAL: NCT04100434
Title: Effect of Evolocumab Added to Moderate-Intensity Statin Therapy on LDL-C Lowering and Cardiovascular Adverse Events in Patients With Acute Coronary Syndrome
Acronym: EMSIACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Chest Hospital (Other)
Responsible Party: Principal Investigator, Yin Liu,MD, Director of coronary care unit, Tianjin Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMSIACS
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Acute Coronary Syndrome; Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor
Keywords: Acute Coronary Syndrome; Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor; Lipid-lowering Drug; Major Cardiovascular Adverse Events
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- the evolocumab plus statin therapy (Experimental): Patients with ACS are treated with atorvastatin (20mg) daily and evolocumab (140 mg) every two weeks throughout the study period
  Interventions: Drug: Evolocumab
- the statin alone therapy (No Intervention): Patients with ACS are treated with atorvastatin (20mg) daily throughout the study period.

INTERVENTIONS:
Drug: Evolocumab — Patients were randomly assigned of the ratio of 1:1 using a computer-generated random number and divided into two treatment groups: the statin alone therapy and the evolocumab plus statin therapy.
  Arms: the evolocumab plus statin therapy

SUMMARY:
The study is an open-label, multicenter, and randomized study(five hospitals).The purpose of this study is to assess the differences in the effects of the evolocumab added to moderate-intensity statin therapy and the moderate-intensity statin only therapy on the regulation of LDL-C levels in patients with acute phase acute coronary syndrome after four weeks of treatment. The primary outcome is the percentage change in LDL-C in weeks 4 and week 12 after treatment. The secondary outcome is the occurrence of MACE after 12 weeks and 1 year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recent hospitalization for acute coronary syndrome: Complies with the diagnostic criteria for acute coronary syndrome (non-ST-segment elevation myocardial infarction, acute ST-segment elevation myocardial infarction, and unstable angina within 72 hours of onset)
* LDL-C level (meet one of the following conditions):

  1. Prior to the study, patients who received intensive statins for more than 4 weeks (the same dose of statin therapy has been sustained for the past four weeks) with LDL-C levels ≥70 mg/dL (≥1.8 mmol/L) or non-HDL-C ≥100 mg /dL (≥2.6mmol/L) are included in the study;
  2. Prior to the study, patients who received moderate-intensity statin therapy for more than 4 weeks (the same dose of statin therapy has been sustained for the past four weeks) with LDL-C levels ≥90 mg/dL (≥2.3 mmol/L) or non-HDL-C≥ 120mg/dL (≥3.1mmol/L) are included in the study;
  3. Prior to the study, patients who do not receive statin therapy or who do not continue to receive statin with LDL-C ≥ 125 mg/dL (≥ 3.2 mmol/L) or non-HDL-C ≥ 155 mg/dL (≥ 4.0 mmol/L).
* Being able to understand research requirements and sign informed consent

Exclusion Criteria:

* Unstable clinical status (hemodynamics or ECG instability)
* Uncontrolled arrhythmia, defined as recurrent or symptomatic ventricular tachycardia and atrial fibrillation with rapid ventricular reaction that the drug cannot control within three months prior to screening
* Severe renal insufficiency, defined as estimated glomerular filtration rate<30ml/min/1.73m2
* Active liver disease or liver dysfunction, whether it is on the patient's medical record or defined as an increase in alanine aminotransferase or aspartate aminotransferase more than 3 times above the upper limit of normal
* Records on statin or rosuvastatin (any dose) intolerance or other statin intolerance
* Known allergies to contrast agents, heparin, aspirin, ticagrelor or clopidogrel
* Known allergies to the supplements required for the use of the drug
* Patients who have been treated with evolocumab or other PCSK9 inhibitors
* Received cholesterol ester transfer protein inhibitors treatment 12 months prior to screening
* Received systemic steroid or cyclosporine treatment in the past 3 months
* Known infections, hemorrhages, metabolic or endocrine disorders as determined by the researchers
* Patients who have been included in other studies
* Patients with active malignant tumor in need of treatment
* Women with fertility (age <50 years, menstruation in the past 12 months), did not receive tubal ligation, oophorectomy or hysterectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in LDL-C | 4 weeks

SECONDARY OUTCOMES:
Major cardiovascular adverse events | 4 weeks and 1 year
  Coronary heart disease death，nonfatal myocardial infarction，hospitalization for unstable angina，unplanned coronary revascularization, and stroke

OTHER OUTCOMES:
The mean percentage change from baseline in LDL-C levels | within 1 year
The proportion of patients with LDL-C <70 mg/dL during treatment | week 4 and week 12
the quality of life of patients | week 12 and week 48
  using EQ-5D-3L questionnaire score to assess the quality of life
The effect of evolocumab on platelet function based on the area under curve | from baseline to 72 hours and baseline to week 4
  using Col/ADP test to evaluate platelet function
the effect of evolocumab on the percentage change of inflammatory markers (high-sensitivity C-reactive protein) | from baseline to week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Chest Hospital,, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jing A, Wang J, Zhang M, Liang Y, Liu J, Zhang N, Wang J, Li X, Li C, Cui Z, Liu Y, Gao J. Effect of PCSK9 inhibitors on the quality of life in patients with acute coronary syndromes - exploratory analysis of the EMSIACS trial. Sci Rep. 2025 Nov 27;15(1):42493. doi: 10.1038/s41598-025-26495-y. PMID 41309899
- [Derived] Gao J, Liu JY, Lu PJ, Xiao JY, Gao MD, Li CP, Cui Z, Liu Y. Effects of Evolocumab Added to Moderate-Intensity Statin Therapy in Chinese Patients With Acute Coronary Syndrome: The EMSIACS Trial Study Protocol. Front Physiol. 2021 Nov 23;12:750872. doi: 10.3389/fphys.2021.750872. eCollection 2021. PMID 34887772